CLINICAL TRIAL: NCT04130451
Title: Efficacy, Safety and Re-occurrence of Pneumothorax and Hydro-pneumothorax With Talc and Pyodine Pleurodesis: A Randomized Control Trial
Brief Title: Efficacy, Safety and Re-occurrence of Pneumothorax and Hydro-pneumothorax With Talc and Pyodine Pleurodesis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Mateen Ahmed Khan, principal investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAKhan
Record Dates: First submitted 2019-09-23; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Secondary Pneumothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre pleurodesis Procedure Fever Pulse rate Respiratory rate Pa (Active Comparator): Pre pleurodesis Fever Pulse rate Respiratory rate Pain thresholds total leukocytes procedure 24 hours before 16 hours before 8 hours before
  Interventions: Drug: PYODINE AND TALC SLURRY
- After Pleurodesis procedure Fever Pulse rate Respiratory rate (Active Comparator): Post pleurodesis Fever Pulse rate Respiratory rate Pain thresholds total leukocytes procdure 24 hours before 16 hours before 8 hours before
  Interventions: Drug: PYODINE AND TALC SLURRY

INTERVENTIONS:
Drug: PYODINE AND TALC SLURRY — pyodine Povidone-iodine is a broad spectrum antiseptic for topical application in the treatment and prevention of wound infection. It may be used in first aid for minor cuts, grazes, burns, abrasions and blisters.
  TALC a white, grey, or pale green soft mineral with a greasy feel, occurring as translucent masses or laminae and consisting of hydrated magnesium silicate

SUMMARY:
Abstract:

INTRODUCTION:

Pneumothorax and hydro-pneumothorax are the most common thoracic injuries and poses a risk of serious morbidity.To prevent the lung from collapsing in such condition, pleurodesis procedure is performed either with surgical pleurodesis,or chemical pleurodesis which adheres outside the lung to the inside chest cavity. The common chemicals that are used are bleomycin, tetracycline, minocycline, slurry of talc and povidoneiodine.

In developed countries, the most common chemical agent used is talc, tetracycline derivatives and bleomycin. However, its clinical results depend on the level of collapse of the lung on the affected side.Internationally, for spontaneous pneumothoraces, talc is the best chemical for pleurodesis procedure which is insufflation through thoracoscopy. However its safety is debateable especially in acute respiratory disease after its administrationwhich made it null and vide consequently. Secondly, in developing countries,medical grade talc availability and affordability remains a constraint. The other suitable chemical is Iodopovidone which is inexpensive and widely used as topical antiseptic in many countries. It also hasshown a safe and effective chemical agent for pleurodesis procedure.

OBJECTIVES:

To determine the efficacy, safety and reoccurrence rate of in pneumothorax and hydro-pneumothorax patients after procedure with talc and pyodine pleurodesis: A comparative study.

MATERIALS AND METHOD:

On the basis of inclusion criteria, the selected 104 patients will be grouped (talc and pyodine) through Non probability, purposive sampling method. In each group 52 willing participants will be included without considering the size of pneumothorax. Six readings of each individual participant will be taken (3 before procedure and 3 after procedure for each group) for pulse and respiratory rate, fever, and total counts of leukocyte. Pain will be assessed on analogue scale. The readings will be taken with 8 hours gap apart. Re-occurrence will be determined after 6 months period of the procedure along with complications if any. The results of both groups will be compared for Efficacy, Safety and Re-occurrence of Pneumothorax and Hydro-pneumothorax.

KEYWORDS:

Pyodine pleurodesis, Talc, hydro-pneumothorax, iodopovidone, pleural effusion, pneumothorax, malignant/prevention & control; Pleurodesis/methods; Recurrence

DETAILED DESCRIPTION:
Introduction:

Pneumothorax and hydro-pneumothorax are the common thoracic injuries which have a severe risk of morbidity. In such a condition either gas or air remains in pleural cavity, a space between visceral and parietal pleura of lung1or air and fluid both are present where air fluid level can be seen in upright chest x-ray of the patient2. To prevent the lung from collapsing in such condition, pleurodesis procedure is performed with surgical or chemical agents which adheres outside the lung to the inside chest cavity1. In surgical pleurodesis, removal of the parietal pleura is done which is an effective way of getting stable pleurodesis. In chemical pleurodesis, the space between the parietal and visceral layer is closed through chemical to prevent further accumulation of fluid. The common chemicals that are used are bleomycin, tetracycline, minocycline, slurry of talc and povidoneiodine

Rational of the study:

There is a little local knowledge is available for use of pyodine which is as effective as talc. If it is determined then it could be easily used in rural areas of the country with a safety involvement. Through determining the efficacy, safety and reoccurrence of pyodine in compare with talc pleurodesis procedure in pneumothorax and hydro-pneumothorax, in patients accordance with systemic inflammatory response syndrome. If the safety, efficacy and less rate of reoccurrence of pyodine are determined as compared to gold standard talc, it will be help fill in treating patients at a remote area where the facility of talc is not available. (Talc chemical lost its validity within 24 hours)

Objective:

To determine the efficacy, safety and reoccurrence rate of Pyodine compared with talc pleurodesis inpatients with pneumothorax.

Hypothesis:

Null Hypothesis:

Talc pleurodesis is more safe having less chances of reoccurring in pneumothorax patients compared to pyodine pleurodesis.

Alternate hypothesis:

Pyodine pleurodesis is as safe, low cost, and easily available with less chances of reoccurring in pneumothorax patients compared to Talc pleurodesis.

METHODS AND MATERIALS:

Study Duration:

Nine months after the approval of synopsis (October 2019 to March 2020)

Study design:

Randomize control trail

Sampling Method:

Non-probability, purposive sampling method

Study setting:

Medical Unit 3, civil hospital, Karachi

Study Instruments:

Structured questionnaire for data collection see in Appendix A

Sample size:

Using sensitivity and specificity in studies (Dr Lin Naing), confidence level 95%, with margin of error 0.05, sample size of the study will be 104 cases divided equally in two groups' i.e.52 in each group.

Data collection procedure:

Study will be conducted after approval of synopsis from Institutional Review Board (IRB), of Dow University of Health Sciences. A written informed consent will also be taken from the participants to put them on Talc or Pyodine group. All patients fulfilling the inclusion criteria will be placed through non probability purposive sampling in groups for pyodine and talc pleurodesis. From all selected patients, 3 readings for pulse and respiratory rate, fever and total leukocyte count for 24 hours at a gap of 8 hours will be recorded prior to procedure. Pain threshold will be determined through visual analogue score 0 to 10 grade. During procedure, it will be assured that bubbling has stopped and lung has expanded. In case of hydro-pneumothorax, the fluid is less 100 ml. After that chest tube pipe will be raise upper the bed level. Than two ampoules of xylocaine injection and 40 ml of 0.9 % saline will be taken. After one or two min, already prepared talc slurry will be instilled in chest tube. In patients selected for pyodine, 40 ml pyodine and 20 ml 0.9% saline will be inserted slowly in chest tube slowly. The patient's tube will remain raised for four to six hours from bed level. After procedure, readings for fever, pulse rate, respiratory rate, and pain threshold of patient with repeated readings with 8 hour gap for 24 hour will be recorded. After repeat chest x-ray, tube will be taken out. Reading of total leukocyte count will be taken after 24 hours of pleurodesis. Follow up will be done for 6 months and reoccurrence rate will be calculated after six month with repeating chest x-ray. Failure of pleurodesis will be determined and put in the result. All the readings will be recorded on the proforma.

Data analysis plan:

The data collected on proforma will be entered in SPSS version 21.0. For each group data, Mean ± SD will be calculated and statistical significance will be determined through independent sample T-Test for quantitative variables like age, pulse and respiratory rate, fever, and total leukocyte count. The pain scores will be determined. The before and after procedure readings in both groups will be analyzed and sensitivity and specificity of pyodine will be determined for with Talc as a gold standard. For qualitative data kike gender, pain score, percentage and frequency will be determined. Confounding and biases will be controlled through strict follow of inclusion criteria.

Ethical Issues:

The ethical approval will be taken from the IRB of Dow University of Health Science, Karachi. A written informed consent will also be taken from the individual participants. The information so collected will be kept in lock and key and nobody other than the researcher and his supervisor will be reached to the data. Right of with draw from the study will be given to all participated patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sex with aged 18 years to 60 years suffering with Pneumothorax and hydro-pneumothorax with lung expanded in chest x-ray.
* Patients of Hydro-pneumothorax with fluid less than 50 ml /24 hour
* Patients having chest tube placed and their column is moving

Exclusion Criteria:

* Patients with broncho-pulmonary fistula will not be a pleurodesis
* Patients with malignant pleural effusion
* Patients with thoraco-scopic procedure having done pleurodesis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2019-10-25 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
fever | 3 months
  it will be measured by thermometer scale and will show the efficacy of the agent as slight fever will show good result because of inflammation.It will show that pleurodesis has been successful and the chemical agent has adherent the two pleural surfaces
pulse rate | 3 months
  according to systemic inflammatory response syndrome, any inflammation can cause increase in pulse rate but tachycardia can occur due to side effects, so pulse rate will show the effectiveness of agent
respiratory rate | 3 months
  it shows how much effective can be the chemical according to systemic inflammatory response syndrome
total leukocyte count | 3 month
  it will show the protocol of systemic inflammatory response syndrome as total leukocyte count can rise in inflammation

OTHER OUTCOMES:
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME | 3 months
  the occurrence of at least two of the following criteria: fever >38.0°C or hypothermia <36.0°C tachycardia >90 beats/minute tachypnea >20 breaths/minute leucocytosis >12*109/l or leucopoenia <4*109/l [1,2

CONTACTS AND LOCATIONS:
Locations (1):
- Mateen Ahmed Khan, Karachi, Pakistan